CLINICAL TRIAL: NCT00191581
Title: Comparison of 2-Hour Postprandial Blood Glucose Excursion in Response to a Standard Test Meal in Insulin-Requiring Diabetic Patients Treated Twice Daily With Either Insulin Lispro Mix 50/50 or Human Insulin Mix 50/50
Brief Title: Local Registration Trial in China Humalog Mix 50
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 9537; F3Z-MC-IOOR
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2006-07-31 (Estimated); Status verified 2006-07

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — isophane insulin, insulin lispro drug combination 50:50

INTERVENTIONS:
Drug: Humalog Mix 50
Drug: Human Insulin Mix 50:50

SUMMARY:
The primary objective of this study is to compare the 2-hour PPBG excursion following a standard test meal in insulin-requiring diabetic patients treated twice daily with human insulin mix 50/50, versus the 2-hour PPBG excursion in patients treated twice daily with insulin lispro mix 50/50.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women who have had either type 1 or type 2 diabetes (World Health Organization[WHO]classification)for at least 2 months and are between the ages of 18 and 70 (inclusive) at the signing of the informed consent.
2. Have been treated with commercially available human insulin mix 50/50 or human insulin mix 30/70 twice daily as the only pharmacological treatment for their diabetes for at least 2 months prior to entering the study.
3. Have an HbA1c between 1.1 and 1.7 times the upper limit of the normal reference rang(inclusive) as determined by a local laboratory within 2 weeks prior to or at Visit 1.
4. Have achieved compliance with their diets and insulin therapies as determined by the investigators and perform regular blood glucose monitoring.
5. Have given informed consent to participate in this study in accordance with local regulations.

Exclusion Criteria:

{1] Have used oral antidiabetic agents, including biguanides, sulfonylureas, glucosidase inhibitors, and insulin-sensitivity enhancers within 30 days prior to entry into the study.

[2] Receive a total daily dose of insulin >2 units/kg.

[3] Have had more than two episodes of severe hypoglycemia (defined as requiring assistance of another person due to disabling hypoglycemia) within 6 months prior to entry into the study.

[4] Have a body mass index >35 kg/m2.

[5] Have serum creatinine > the upper limit of normal (ULN), as determined by a local laboratory.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2005-03; Study Completion 2006-04

PRIMARY OUTCOMES:
The primary objective of this study is to compare the 2-hour PPBG excursion following a standard test meal in IDDM patients treated BID with human insulin mix 50/50, vs the 2-hour PPBG excursion in patients treated BID with insulin lispro mix 50/50

SECONDARY OUTCOMES:
The secondary objectives of the study are:
Assess hemoglobin A1c (HbA1c) values at baseline and after treatment with insulin lispro mix 50/50.
Assess HbA1c values at baseline and after treatment with human insulin mix 50/50.
To compare human insulin mix 50/50 with insulin lispro mix 50/50 with regard to
Effects on HbA1c values obtained at the end of each treatment period;
Effects on fasting blood glucose values obtained throughout the study;

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST, Study Director — Eli Lilly and Company
Locations (2):
- China (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Beijing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Guangzhou

REFERENCES:
- [Derived] Gao Y, Li G, Li Y, Guo X, Yuan G, Gong Q, Yan L, Zheng Y, Zhang J. Postprandial blood glucose response to a standard test meal in insulin-requiring patients with diabetes treated with insulin lispro mix 50 or human insulin mix 50. Int J Clin Pract. 2008 Sep;62(9):1344-51. doi: 10.1111/j.1742-1241.2008.01850.x. Epub 2008 Jul 24. PMID 18657196